CLINICAL TRIAL: NCT07266896
Title: Patient-specific Finite Element Analysis of Immediate Loading in the Edentulous Maxilla: Comparison of Three Implant Configurations Using Digital Twins.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Odonto07
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atrophic Edentulous Maxilla
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: numerical study — CBTS Scans (Cone Beam Computed Tomography) perform as part of routine care

SUMMARY:
Rehabilitation of severely atrophic edentulous maxillae with dental implants pose a significant clinical challenge. Immediate loading in grafted bone is often debated due to concerns about stress distribution and osseointegration. This study aimed to compare stress distribution in the maxilla using three full-arch implant configurations-all-on-four, all-on-six, and quad-zygomatic implants-in a single patient, to determine the safest and most favorable approach for immediate loading in grafted bone. Two CBCT scans from a 64-year-old female patient, before and after bone grafting (allograft with onlay grafting and sinus augmentation), were used to generate three patient-specific finite element models. Each model included the maxilla, implants in the respective configuration, abutments, and a full-arch prosthesis. Von Mises stresses in cortical and cancellous bone, implants, abutments, and prosthesis, as well as maximum bone displacement, were analyzed. Our results demonstrated that the all-on-six configuration provided the most favorable biomechanical outcome, with homogeneous cortical stress distribution, reduced stress in implants and prosthesis, and bone displacement fully compatible with immediate loading in grafted bone. The all-on-four model showed stress peaks at tilted abutments and cantilevers, whereas the quad-zygomatic model distributed implant and abutment stresses efficiently but induced higher cortical bone stresses, still within physiological limits.This patient-specific digital twin study demonstrates that immediate loading in full-arch grafted bone is biomechanically safe and optimal, with the all-on-six configuration providing superior stress distribution. These findings support clinical decision-making for immediate loading protocols and highlight the value of patient-specific FEA in planning complex maxillary rehabilitations.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous maxillae, have had full-arch bone reconstruction

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Edentulous maxillae, have had full-arch bone reconstruction in order to use the scanner before the bone graft and the scanner after the bone graft and simulate two configurations (all on four and quad zygomatic) on the digital model from the first scanner, and one implant configuration (all on six) on the digital model from the second scanner.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Stress distribution in the Maxillary Bone | At inclusion
  Finite element analysis (FEA) a numerical simulation method that models how mechanical forces affect anatomical structures. This technique visualizes stress, tension, compression and displacement zones in the maxillary bone. Stress values are expressed in megapascals (MPa) and displacements in microns (μm).
Stress distribution in the Implants | At inclusion
  Finite element analysis (FEA). This technique visualizes stress, tension, compression and displacement zones in the implant. Stress values are expressed in megapascals (MPa) and displacements in microns (μm).
Stress distribution in the Prosthesis | At inclusion
  Finite element analysis (FEA). This technique visualizes stress, tension, compression and displacement zones in the prosthesis. Stress values are expressed in megapascals (MPa) and displacements in microns (μm).

SECONDARY OUTCOMES:
Accuracy of the digital model digital twin of real patient | At inclusion
  Scan of his edentulous maxilla

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France